**Official Title**: Transmeridian Travel in Elite Female Athletes: Efficacy of Maintaining a Home-Based Schedule to Optimize Sleep & Performance

**NCT #**: NCT06920225

**Document Date**: 18 August 2025

**Title of research study:** Transmeridian Travel in Elite Female Athletes: Efficacy of Maintaining a Home-Based Schedule to Optimize Sleep & Performance

**Investigator:** Timothy Griest, PhD(c)

Faculty Advisor: Dr. Michael Ormsbee, PhD; Director, Institute of Sports Sciences & Medicine

**<u>Key Information</u>**: The following is a short summary of this study to help you decide whether or not to be a part of this study. More detailed information is listed later on in this form.

#### Why am I being invited to take part in a research study?

We invite you to take part in a research study to determine if maintaining an East Coast time zone schedule during West Coast travel will help sleep and performance.

#### What should I know about a research study?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

#### Why is this research being done?

The purpose of this study is to determine if maintaining an East Coast time zone schedule during West Coast travel will help objective and subjective sleep and physical performance.

Jet lag that occurs after traveling across time zones can negatively impact both sleep and physical performance, lowering the team's chances of winning their competitions. Optimizing performance and recovery is important for athletic success, and this strategy could help with that during away competitions.

# How long will the research last and what will I need to do?

We expect that you will be in this research study for  $\sim$ 36 days, across the span of  $\sim$ 2-3 months throughout the competition season.

The first visit will include receiving this informed consent and screening questionnaires (medical, sleep, chronotype, and menstrual history). We will obtain DEXA information from your previous scans. The remaining visits will occur throughout the competition season. We will be assessing sleep and physical performance for 3 days before and the days of (~5 days) four different series of games. The four series will include one home series, one road series on the East Coast, and two road series on the West Coast. During one of the West Coast series, you will maintain an East Coast time zone schedule, while during the other trip you will transition to a West Coast time zone schedule. Before, and during each series, you will be asked to wear your WHOOP band as much as possible so that we can get objective sleep quality and recovery data. We will also ask you to complete a short survey in the morning of these days to assess your subjective sleep quality and recovery. Finally, you will perform countermovement jumps on the force plates, grip strength testing, and reaction time testing once ~2 days before the series and once before each of the games. The study design is illustrated in Figure 1.



Figure 1. Study Design

More detailed information about the study procedures can be found under "What happens if I say yes, I want to be in this research?"

### Is there any way being in this study could be bad for me?

There is a small risk of acute muscle or bone injuries from countermovement jumps and grip strength testing; however, this risk is low.

More detailed information about the risks of this study can be found under "Is there any way being in this study could be bad for me? (Detailed Risks)"

### Will being in this study help me in any way?

We can't guarantee that participating in this research will have specific benefits for you or anyone else. However, possible benefits include learning about a strategy that may help optimize sleep and performance during travel across multiple time zones.

### What happens if I do not want to be in this research?

Participation in research is completely voluntary. You can decide to participate or not to participate. Your alternative to participating in this research study is to not participate. Refusal to participate will involve no penalty or loss of benefits to which you are entitled.

**<u>Detailed Information:</u>** The following is more detailed information about this study in addition to the information listed above.

#### Who can I talk to?

If you have questions, concerns, or complaints, or have experienced a research-related injury or think that the research has hurt you, contact the research team at:

Tim Griest (717) 466-4286 Tdg21c@fsu.edu

This research has been reviewed and approved by an Institutional Review Board ("IRB"). You may talk to them at 850-644-7900 or humansubjects@fsu.edu if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

### How many people will be studied?

We expect about 18 people will be in this research study.

## What happens if I say "yes" to being in this research?

#### **Initial Visit: (~60 minutes)**

We will meet with you at one of the meeting rooms in your facility to complete informed consent and the initial screening forms. The screening forms include the following: Past Medical History, Menstrual Status, Sleep History, and Chronotype questionnaire.

#### **Baseline Days and Nights (PRE3-PRE1)**

Each morning you will complete a short sleep survey. We request you complete this 30-60 minute after waking up. You will receive a reminder in the morning to complete this survey. We also request that you wear your WHOOP band each of these nights. We will collect the WHOOP data from each morning through a representative at WHOOP. During one of the days (PRE2), you will perform the physical testing, including countermovement jumps, grip strength testing, and reaction time testing.

#### **Competition Days and Nights (COMP1-COMP5)**

Each morning you will complete a short sleep survey. We request you complete this 30-60 minute after waking up. You will receive a reminder in the morning to complete this survey. We also request that you wear your WHOOP band each of these nights. We will collect the WHOOP data from each morning through a representative at WHOOP. During each of these

days, you will perform the physical testing, including countermovement jumps, grip strength testing, and reaction time testing.

The above process (Baseline & Competition) will be repeated four times, once during a home series, once during an away series on the East Coast, and twice during an away series on the West Coast. During one of the West Coast series, you will maintain an East Coast time zone schedule, while during the other trip you will transition to a West Coast time zone schedule.

### What are my responsibilities if I take part in this research?

If you take part in this research, you will be responsible to complete the sleep surveys, wear your WHOOP band, and complete the physical testing sessions with maximum effort. You will also be responsible to download the Sway Medical application and complete the tests to the best of your ability.

## What happens if I say "yes," but I change my mind later?

You can leave the research at any time, it will not be held against you. If you decide to leave the research, contact the investigator so that the investigator can ensure you don't receive any more notifications about the study. If you choose to leave the research at any time, there will be no penalty or loss of benefits to which you are otherwise entitled.

## Is there any way being in this study could be bad for me? (Detailed Risks)

The risks of this study are not significantly different than the risks you face on a daily basis as an athlete at Florida State University.

**Physical Risks:** Although the risk is small, performing countermovement jumps and grip strength testing can but too much strain on the body and cause injury. Since these movements are ones that are often performed in your training programs, the risk of injury is decreased. You will also be supervised during each of these testing sessions, decreasing the risk even more.

**Psychological Risks:** Although the risk is small, the surveys may be a slight inconvenience due to the time they take to complete. We have decreased this risk by making sure we have the smallest number of questions we need to answer our questions. The use of an electronic software will also speed up this process

There are no known or expected privacy, legal, social, or economic risks.

You and your insurance company will be charged for the health care services that you would ordinarily be responsible to pay. In some cases, insurance will not pay for services ordinarily covered because these services were performed in a research study. You should check with your insurance to see what services will be covered by your insurance and what you will be responsible to pay.

## What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information. However, we cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB and other representatives of this organization.

If identifiers are removed from your identifiable private information or identifiable samples that are collected during this research, that information or those samples could be used for future research

studies or distributed to another investigator for future research studies without your additional informed consent.

We may publish the results of this research. However, we will keep your name and other identifying information confidential to the extent allowed by law.

### Can I be removed from the research without my OK?

The person in charge of the research study or the sponsor can remove you from the research study without your approval. Possible reasons for removal include:

- Failure to complete > 90% of the daily subjective sleep surveys
- Failure to wear WHOOP device for > 95% of study intervention nights
- Failure to complete any of the physical performance testing sessions

We will tell you about any new information that may affect your health, welfare, or choice to stay in the research.

#### What else do I need to know?

If you need medical care because of taking part in this research study, contact the investigator and medical care will be made available. Generally, this care will be billed to you, your insurance, or other third party. Florida State University has no program to pay for medical care for research-related injury.

Upon successful completion of each condition, you will be provided with a complementary \$50 VISA gift card for your time and effort. The gift card will be delivered by the PI and/or the research team after completion of the study.

## **Signature Block for Capable Adult**

Your signature documents your permission to take part in this research.

| Signature of subject | Date |
|---------------------------------------|----------|
| Printed name of subject | <u> </u> |
| Signature of person obtaining consent | Date |

| Permission to Take Part in a Human Research Study |
|---------------------------------------------------|